CLINICAL TRIAL: NCT00273533
Title: Effects of Ramipril on Endothelial Function in Patients With Rheumatoid Arthritis
Brief Title: Ramipril in Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Sanofi (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: HOE498/6007
Record Dates: First submitted 2006-01-06; First posted 2006-01-09 (Estimated); Last update posted 2008-07-22 (Estimated); Status verified 2006-10

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Ramipril

INTERVENTIONS:
Drug: Ramipril

SUMMARY:
The present study is designed to evaluate the hypothesis that the Angiotensin-Converting Enzyme (ACE) inhibitor Ramipril improves vascular function and reduces markers of low-grade chronic inflammation and oxidative stress in patients with Rheumatoid Arthritis.

DETAILED DESCRIPTION:
The effect of an 8-week treatment with either ramipril or placebo is studied using a randomized, double-blind, and crossover protocol. After given written informed consent, baseline characteristics including physical examination, ECG, blood sample and a noninvasive assessment of endothelial function are obtained. The patients are randomly assigned to receive either ramipril 10mg (up-titration-scheme: starting with 2.5mg in Week1, then 5mg in Week2 followed by 2-5mg for the final 6 weeks) followed by placebo or vice versa.The individual disease-modifying antirheumatic drug therapy is continued throughout the study. The examinations are repeated after 8 weeks treatment of the first and 8 weeks after the second study drug. At week 1 and 2 in each treatment period a safety visit is scheduled.

ELIGIBILITY:
Inclusion Criteria:

* patients with rheumatoid arthritis (4 out of 7 ARA criteria must be fulfilled to establish diagnosis) on stable background therapy for the last three months
* endothelial dysfunction (FMD < 4%, FMD:Flow-Mediated-Dilatation)
* non-smokers

Exclusion Criteria:

* previous myocardial infarction, coronary intervention or coronary surgery
* previous treatment with statins in the last 6 months
* previous treatment with ACE-inhibitors in the last 6 months
* uncontrolled hypertension SAP/DAP > 160/90 mmHg (SAP:Systolic Arterial Pressure, DAP:Diastolic Arterial Pressure)
* dyslipidemia (LDL-cholesterol > 4.9 mmol)
* normal CRP < 3 mg/l
* overweight BMI > 35kg/m2
* anaemia (hemoglobin < 10g/dl)
* kidney disease (creatinine > 150 umol/l)
* insulin-dependent diabetes mellitus
* congestive heart failure (> NYHA I)
* AV-Block>I
* pregnancy
* angio-edema
* malignancy or chronic infection
* drug abuse

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2004-06; Study Completion 2006-07

PRIMARY OUTCOMES:
Endothelial dysfunction evaluated on weeks 8 and 16.

SECONDARY OUTCOMES:
Alteration of inflammatory parameters: C-reactive Protein, TNFa, Interleukin 6 on weeks 8 and 16.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Shokry, Study Director — Sanofi

REFERENCES:
- [Derived] Flammer AJ, Sudano I, Hermann F, Gay S, Forster A, Neidhart M, Kunzler P, Enseleit F, Periat D, Hermann M, Nussberger J, Luscher TF, Corti R, Noll G, Ruschitzka F. Angiotensin-converting enzyme inhibition improves vascular function in rheumatoid arthritis. Circulation. 2008 Apr 29;117(17):2262-9. doi: 10.1161/CIRCULATIONAHA.107.734384. Epub 2008 Apr 21. PMID 18427133